CLINICAL TRIAL: NCT01320319
Title: Effect of EPA Nutritional Supplementation on Markers of Aerobic Performance, Lean Muscle Mass and Quality of Life on Patients Undergoing Curative Resection of Colorectal Cancer
Brief Title: Effect of EPA on Aerobic Performance, Muscle, and Quality of Life in Colorectal Cancer Surgery Patients
Acronym: EPA-colo
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11005
Record Dates: First submitted 2011-03-02; First posted 2011-03-22 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Nutritional Supplementation with EPA (Experimental): This arm will receive the nutritional supplementation of EPA 960mg Three times a day.
  Interventions: Dietary Supplement: Experimental: Nutritional Supplementation with EPA

INTERVENTIONS:
Other: Placebo — Capsule form, 960 mg to be taken three times a day.
  Arms: Placebo
Dietary Supplement: Experimental: Nutritional Supplementation with EPA — Capsule form, EPA, 960mg to be taken three times a day.
  Arms: Nutritional Supplementation with EPA

SUMMARY:
Primary Aim is to test the Hypothesis: Nutritional supplementation with 960mg EPA three times a day positively affects muscle function and mass (assessed by muscle biopsies, assays of cellular aerobic function and DEXA scan) and inflammation (measuring cellular markers of inflammation) in patients undergoing resection of colorectal cancers.

The secondary aim is to evaluate aerobic performance assessed by cardiopulmonary exercise testing (CPEX) and perioperative outcome in patients with colorectal cancer post surgical resection.

DETAILED DESCRIPTION:
Cancer is well documented to cause weight loss and cachexia (1). An inflammatory process driven by the presence of a tumour, can result in reduced food intake (2), increased metabolic output (3) and loss of skeletal muscle (1). They have reduced fitness and feeling of lethargy that affects activities of daily living and quality of life. The process explaining this is not well understood but thought to be due to diminished skeletal muscle mass and performance. When cancer patients undergo surgery, the trauma of surgery, entails an inflammatory process that furthermore leads to more of the above (4). Reducing this inflammatory insult would positively impact fitness, ability to respond to infections, affect length of stay in hospital, recovery from surgery and quality of life following surgery.

Eicosapentaenoic acid (EPA) is an omega-3-fatty acid, derived from fish oil and a commonly available nutritional supplement. It is believed to reduce the inflammatory effect of cancer and the trauma of surgery, in turn dampening the catabolic effect causing skeletal muscle loss. Studies on oesophageal cancer patients have previously suggested that EPA can preserve lean muscle mass (5). The investigators expect EPA to cause less lean muscle loss and improved aerobic performance. High dietary intake is not thought to have health risks (6) and EPA has recently been trialed in infant milk formulas with no adverse effects (7).

The investigators plan to recruit patients from colorectal clinic, who are due to have surgery for colorectal cancer, and give them EPA or placebo, from 5 days prior to surgery to up to 21 days following surgery. The investigators would like to measure markers of muscle function and inflammation, muscle mass, exercise performance on by cardiopulmonary exercise testing, muscle biopsy and muscle grip strength on a dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients listed for open curative tumour resection by means of: Right Hemi Colectomy, Left Hemi-colectomy or Anterior Resection, not having neo-adjuvant chemotherapy.
* Aged 18 - 85 years old.

Exclusion Criteria:

* Strenuous exercise 48 hours before the preoperative assessment.
* Intramuscular injections within 48 hours of any study day.
* Known peripheral neuropathy or myopathy.
* Patients with mobility problems, wheelchair bound or have suffered a previous cerebro-vascular accident with residual impairment of mobility.
* Patients with major/ minor trauma (Motor vehicle accidents or ground falls, firearm injury, drowning, struck by and against injuries).
* Pregnant women. Pregnancy test will be done at the beginning of the study day.
* Patients without mental capacity to give signed consent.
* Patients already taking fish-oil derived nutritional supplement.
* Patients with impaired oral intake.
* Patients known to have metastatic disease.
* Patients having neoadjuvant chemotherapy prior to resection, which may confound results.
* Patients having laparoscopic procedures.
* Patients identified having cardiorespiratory comorbidity considered unsuitable for surgery: unstable angina, myocardial infarction within last 3 months, severe aortic stenosis, pulmonary hypertension, HOCM, acute myopericarditis, chronic heart failure New York Heart Association class 3 and above and impaired left ventricular ejection fraction (less than 43%). Respiratory contraindications include severe COPD, emphysema, fibrosing alveolitis, Interstitial lung disease and FEV1 less than 1.5.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Nutritional supplementation with 960mg EPA three times a day positively affects muscle function and mass | Baseline and 6 weeks post-op
  Muscle function and mass will be assessed by muscle biopsies, assays of cellular aerobic function and DEXA scan and inflammation (measuring cellular markers of inflammation).

SECONDARY OUTCOMES:
The secondary aim is to look at the aerobic performance. | Baseline and 5 weeks post-op.
  The secondary aim is to look at the aerobic performance assessed by cardiopulmonary exercise testing (CPEX) and perioperative outcome in patients with colorectal cancer post surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, Principal Investigator — University of Nottingham
Locations (1):
- School of Graduate Entry Medicine & Health, Royal Derby Hospital, Derby, Derby, United Kingdom

REFERENCES:
- [Derived] Hossain T, Phillips BE, Doleman B, Lund JN, Williams JP. A double-blind randomized controlled trial of the effects of eicosapentaenoic acid supplementation on muscle inflammation and physical function in patients undergoing colorectal cancer resection. Clin Nutr. 2020 Jul;39(7):2055-2061. doi: 10.1016/j.clnu.2019.09.009. Epub 2019 Oct 11. PMID 31648815